CLINICAL TRIAL: NCT04109482
Title: A Phase 1/2, Open Label, Multicenter Trial to Assess the Safety and Efficacy of MB-102 in Patients With Relapsed or Refractory Blastic Plasmacytoid Dendritic Cell Neoplasm
Brief Title: Trial to Evaluate the Safety and Efficacy of MB-102 in Patients With BPDCN.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business reasons.
Sponsor: Mustang Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MB102-CD123-001
Record Dates: First submitted 2019-09-25; First posted 2019-09-30 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2023-06

CONDITIONS: Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN)
Keywords: CD123 CAR-T; BPDCN; Blastic plasmacytoid dendritic cell neoplasm
MeSH Terms: conditions — Blastic Plasmacytoid Dendritic Cell Neoplasm | interventions — relmapirazin; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Relapsed or Refractory BPDCN (Experimental): Treatment with MB-102.
  Interventions: Biological: MB-102; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: MB-102 — The study drug, MB-102 consists of adoptively transferred T cells that are genetically modified using a self-inactivating (SIN) lentiviral vector to express a CD123-specific, CD28-costimulatory chimeric antigen receptor (CAR) as well as a truncated human epidermal growth factor receptor (EGFRt) (CD123.CD28.CD3ζ.EGFRt+T cells) derived from autologous leukapheresis which is administered after a lymphodepletion regimen.
  Single dose of MB-102 up to 600 x 10 6 CART-T+ cells (Day 0) as defined by Phase 1 will be administered.
  Other Names: CD123 CAR-T
Drug: Fludarabine — Fludarabine 30 mg/m2/day IV (3 days) on days -5, -4, and -3
  * A 20% dose reduction (24 mg/m2/day IV (3 days) on days -5, -4, and -3) is required for patients with moderately impaired renal function (creatine clearance ≤ 70 mL/min).
  Other Names: Fludara
Drug: Cyclophosphamide — Cyclophosphamide 300 - 500 mg/m2/day IV (3 days) on days -5, -4, and -3
  Other Names: Cytoxan

SUMMARY:
A phase 1/2 study to assess the safety and efficacy of MB-102 in patients with relapsed or refractory BPDCN

DETAILED DESCRIPTION:
The Phase 1 portion of the study will determine the maximum tolerated dose of MB-102.

The Phase 2 portion of the trial will evaluate the efficacy of MB-102 in relapsed or refractory BPDCN.

ELIGIBILITY:
Inclusion Criteria:

Blastic Plasmacytoid Dendritic Cell Neoplasm

1. Patients with a diagnosis of BPDCN according to WHO classification (Arber et al., 2016) confirmed by hematopathology and histological/cytological evidence of BPDCN in the peripheral blood, bone marrow, spleen, lymph nodes, skin and/or other sites who have failed one prior therapy.

   General Inclusion Criteria
2. Male and female patients ≥ 18 years of age at the time of consent.
3. Written informed consent in accordance with federal, local, and institutional guidelines.
4. Must be able to adhere to the study visit schedule and other protocol requirements.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Meet the following laboratory criteria:

   * Absolute lymphocyte count (ALC) > 100/mm3
   * ALT/SGPT and AST/SGOT < 2.5x the upper limit of normal (ULN) unless due to underlying disease state
   * Calculated creatinine clearance ≥ 45.0 mL/min as estimated by Cockcroft Gault and dialysis independent
   * Total bilirubin ≤ 3.0 mg/dL

     * Patients with Gilbert's Syndrome must have a total bilirubin < 5.0 mg/dL.
   * Serum albumin ≥ 3.2 g/dL
7. Cardiac ejection fraction ≥ 45%, with no evidence of pericardial effusion as determined by an echocardiogram (ECHO) or if not available, a multigated acquisition scan (MUGA).
8. Females participants of childbearing potential must have a negative serum test.
9. Patients must agree to use a highly effective method of contraception if procreative potential exists from the start of the study until one year after the completion of lymphodepletion for females and 4 months after completion of lymphodepletion for males.
10. Patients with a previously treated malignancy if treatment of that malignancy was completed greater than 2 years before screening and the patient has no evidence of disease at the time of screening.
11. Patients who have previously undergone allogenic or autologous bone marrow transplants are allowed.
12. Centrally confirmed CD-123 positivity on the bone marrow, or for patients without bone marrow involvement local pathology assessments within 28 days from Screening, showing evidence of CD-123 positivity of skin/lymph node biopsy.

Exclusion Criteria:

1. Patients with a corticosteroid dependence on doses greater than physiological replacement i.e., prednisone no more than 7.5 mg/day or hydrocortisone less than 12mg/m2/day.
2. Contraindication or hypersensitivity to fludarabine or cyclophosphamide.
3. Hypersensitivity or known history of allergic reactions attributed to tocilizumab, Cetuximab, or other anti-EGFR -monoclonal antibodies.
4. Immunotherapy treatments within 28 days prior to leukapheresis.
5. Previous treatment with anti-CD123 CAR-T treatment.

   * Previous treatment with non-CAR-T anti-CD123 agents is allowed e.g. tagraxofusp-erzs.
6. Previous treatment with any other antileukemic or investigational agent within 7 days of leukapheresis.

   * Hydroxyurea is allowed up to 3 days prior to leukapheresis.
7. Patients with history or active seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease or any autoimmune disease with CNS involvement.
8. Patients with known CNS leukemic involvement that are refractory to intrathecal chemotherapy and/or cranio-spinal radiation that have NOT been effectively treated to complete remission (defined as < 5 WBC/mm3 and no blasts in CSF).
9. Patients with active Graft versus Host Disease (GVHD).
10. Acute active infection

    * Patients being administered prophylactic antibiotics, antivirals, or antifungals are permitted.
11. Patients who have any form of primary immunodeficiency, such as severe combined immunodeficiency disease, human immunodeficiency virus (HIV), or acquired immune deficiency syndrome (AIDS).
12. Active infection with hepatitis B or C.
13. Patients requiring supplemental oxygen or mechanical ventilation or oxygen saturation < 92% on room air.

    * Patients with an oxygen saturation < 92%, a pulmonary function test with a result of Diffusing capacity of the lungs for carbon monoxide (DLCO) of ≥ 40% of predicted and a forced expiratory volume in one second (FEV1) > 45% predicted will be accepted.
14. Patients with decompensated hepatic cirrhosis/liver failure.
15. Pregnant or lactating females.
16. Any other clinically significant medical disease or condition that, in the investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Phase 1: Safety and Tolerability as measured by the number of patients with treatment related adverse events | 28 Days
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 in Phase 1
Phase 1: Maximum Tolerated Dose (MTD) and recommended Phase 2 dose | 28 Days
  To determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose of MB-102
Phase 2: Response Rate of patients with BPDCN | up to 3 years
  Relapsed or refractory Blastic Plasmacytoid Dendritic Cell Neoplasm is measured by a response rate which consists of Complete Response and clinical Complete Response and Complete Response with incomplete hematologic recovery (CR + CRc + CRi) at day 28 post infusion

SECONDARY OUTCOMES:
Phase 2: BPDCN - DOR | up to 3 years
  Duration of Response
Phase 2: BPDCN - PFS | up to 3 years
  Progression-Free Survival
Phase 2: BPDCN - OS | up to 3 years
  overall survival
Phase 2: BPDCN - MRD | up to 3 years
  CR MRD- Response Rate for patients with CR and CRi
Phase 2 - Adverse events | up to 3 years
  Incidence of treatment-emergent AEs (TEAEs), including SAEs, therapy-related AEs or death.
Phase 2 -Change from Baseline in the European Organization for Research and Treatment (EORTC) QLQ-C 30 Version 3.0. | up to 3 years
  The European Organization for Research and Treatment (EORTC) QLQ-C 30 Version 3.0 is an integrated, modular approach for evaluating the quality of life of patients participating in international clinical trials. The questionnaire is designed to measure cancer patients' physical, psychological and social functions. The questionnaire is composed of 5 multi-item scales (physical, role, social, emotional and cognitive functioning) and 9 single items (pain, fatigue, financial impact, appetite loss, nausea/vomiting, diarrhea, constipation, sleep disturbance and quality of life).
  It utilizes a four-point scales for the first 28 questions which are coded with response categories as "Not at all", "A little", "Quite a bit" and "Very much.". the final two question consist of an overall physical condition questions which have employed a 7-point response scale where the higher number indicates a better overall health.
Phase 2 - Change from Baseline in the Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) Version 4.0. | up to 3 years
  The Functional Assessment of Cancer treatment for cancer, and a transplant-specific module, bone marrow transplant (BMT) concerns, that addresses disease and treatment-related questions specific to BMT.
  It utilizes a 5 point scale assessing physical, social, emotional, functional and other well-being concerns. Response categories are coded as "Not at all", "A little bit", "Somewhat", "Quite a bit" and "Very much.".
Phase 2 - Number of patients showing evidence of replication competent lentivirus | up to 3 years
  To confirm the absence of replication competent lentivirus

CONTACTS AND LOCATIONS:
Overall Officials: Lihua E Budde, MD, Principal Investigator — City of Hope Medical Center
Locations (4):
- United States (4):
  - City of Hope Medical Center, Duarte, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No